CLINICAL TRIAL: NCT04858529
Title: Neoadjuvant TCHP Versus THP in Patients With Human Epidermal Growth Factor Receptor 2-positive Breast Cancer (neoCARHP) : a Randomized, Open-label, Multicenter, Phase III Trial
Brief Title: Neoadjuvant TCHP Versus THP in Patients With HER2-positive Breast Cancer (neoCARHP Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, M.D., Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201101
Record Dates: First submitted 2021-04-18; First posted 2021-04-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neoadjuvant Therapies for HER2+ Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THP (Experimental)
  Interventions: Drug: investigator-selected taxane/trastuzumab/pertuzumab (THP)
- TCHP (Active Comparator)
  Interventions: Drug: investigator-selected taxane/carboplatin/trastuzumab/pertuzumab (TCHP)

INTERVENTIONS:
Drug: investigator-selected taxane/carboplatin/trastuzumab/pertuzumab (TCHP) — investigator-selected taxane/carboplatin/trastuzumab/pertuzumab (TCHP)
  Arms: TCHP
Drug: investigator-selected taxane/trastuzumab/pertuzumab (THP) — investigator-selected taxane/trastuzumab/pertuzumab (THP)
  Arms: THP

SUMMARY:
The neoCARHP study was a randomized, open-label, multicenter, phase III, neoadjuvant trial. This study aimed to compare the efficacy and safety of TCHP with THP neoadjuvant setting for HER2-positive breast cancer. Patients will be randomized at a 1:1 ratio into TCHP or THP, respectively, and will be treated every 3 weeks before surgery.The primary endpoint was the percentage of pCR (ypT0/is, ypN0), which was defined as the absence of any residual invasive cancer in both the breast and axillary lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* To take part in the trial, patients must be aged > 18 years old and supply a signed informed consent form.

Patients must also have breast cancer meeting the following criteria:

* Histologically confirmed invasive breast carcinoma
* Clinical stage II-IIIC at presentation. HER2-positive breast cancer scored as 3+ by immunohistochemistry (IHC) in > 10% of immunoreactive cells, or HER2 gene amplification (ratio of HER2 gene signals to centromere 17 signals ≥2.0) by in situ hybridization (ISH).

Known hormone receptor status (ER and PR). Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1. Completed all necessary baseline laboratory and radiologic examinations prior to randomization.

Baseline left ventricular ejection fraction (LVEF)≥55% measured by echocardiography (ECHO).

Women who are not postmenopausal (≥12 months of amenorrhea) or surgically sterile (absence of ovaries and/or the uterus) must agree to remain abstinent or to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception during the treatment period and for at least 6 months after the last dose of study treatment.

Clinical diagnosis of Alzheimer's Disease. Must be able to swallow tablets. All patients must be able to comply with the study protocol, according to the investigator's judgment.

Exclusion Criteria:

* Stage IV (metastatic) breast cancer Inflammatory breast cancer Previous anti-cancer therapy or radiotherapy for any malignancy. A history of other malignancies, except for carcinoma in situ of the cervix or squamous or basal cell carcinoma.

Concurrent anti-cancer treatment in another clinical trial, including hormone therapy, bisphosphonate therapy, or immunotherapy.

Received a major non-breast cancer-related surgical procedure within the 4 weeks before randomization or from which the patient has not fully recovered.

A serious cardiac illness or medical condition, including but not limited to the following:

Documented history heart failure or systolic dysfunction (LVEF < 50%). High-risk uncontrolled arrhythmia, such as atrial tachycardia with a heart rate >100 bpm at rest, significant ventricular arrhythmia (e.g., ventricular tachycardia), or higher-grade atrioventricular (AV) block (i.e., Mobitz II second-degree AV block or third-degree AV block).

Angina pectoris requiring anti-angina medication. Clinically significant valvular heart disease. Evidence of transmural infarction on ECG Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg) Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness.

Any of the following abnormal laboratory tests immediately prior to randomization:

Total bilirubin > 1.5 × upper limit of normal (ULN) or, for cases of known Gilbert's syndrome, total bilirubin > 2 × ULN Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.25 × ULN Alkaline phosphatase > 2.5 × ULN Serum creatinine > 1.5 × ULN Total white blood cell (WBC) count < 2500 cells/uL Absolute neutrophil count <1500 cells/uL Platelet count <100,000 cells/uL Sensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol Pregnant or lactating: a negative serum pregnancy test is required for all women who are not postmenopausal (≥ 12 months of amenorrhea).

Insulin dependent diabetes. Thyroid disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(ypT0/is,ypN0, pCR) | 18 weeks
  defined as the absence of invasive tumor cells in breast and axilla, ypT0/is ypN0

SECONDARY OUTCOMES:
Clinical response during neoadjuvant therapy | 18 weeks
  Clinical response during neoadjuvant therapy, according to RECIST v1.1.
The percentage of patients who underwent breast-conserving surgery | 18 weeks
Event-free survival (EFS) | until disease progression or recurrence or until 5 years after randomization of the last patient, which ever occurs first.
  Event-free survival (EFS), defined as the time from randomization to the first report of one of the following events:
  1. Disease progression (before surgery), as determined by the investigator according to RECIST v1.1. Any evidence of in situ contralateral disease will not be identified as progressive disease (PD). Any evidence of invasive contralateral disease will be considered as disease progression
  2. Disease recurrence (local, regional, distant, or contralateral) after surgery.
  3. Death from any cause.
Disease-free survival (DFS) | until disease progression or recurrence or until 5 years after randomization of the last patient, which ever occurs first.
  Disease-free survival (DFS), defined as the time from the first date of no disease (i.e., date of surgery) to the first documentation of one of the following events:
  1. Disease recurrence (local, regional, distant, or contralateral) after surgery
  2. Death from any cause
Safety Outcome Measures | until disease progression or recurrence or until 5 years after randomization of the last patient, which ever occurs first.
  The safety outcome measures for this study are the incidence, type, and severity of adverse events and serious adverse events.
Overall survival, defined as the time from randomization to death from any cause. | from randomization to death from any cause.
  Overall survival, defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu T, Huang YH, Li W, Wu CG, Zhang YM, Zheng XX, Zhang TF, Lin YY, Liu ZY, Ye GL, Lin Y, Wu ZY, Wang K. A non-invasive artificial intelligence model for identifying axillary pathological complete response to neoadjuvant chemotherapy in breast cancer: a secondary analysis to multicenter clinical trial. Br J Cancer. 2024 Sep;131(4):692-701. doi: 10.1038/s41416-024-02726-3. Epub 2024 Jun 25. PMID 38918556